CLINICAL TRIAL: NCT04835363
Title: Early Occupational Therapy Intervention in the Hospital Discharge After Stroke: Study Protocol for a Randomized Controlled Trial
Brief Title: Early Occupational Therapy Intervention in the Hospital Discharge After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Patricia García Perez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOTIHDAS2021
Record Dates: First submitted 2021-03-25; First posted 2021-04-08 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: patient discharge; occupational therapy; rehabilitation; caregivers
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group - Patients (No Intervention): Usual care and rehabilitation.
- OT intervention group - Patients (Experimental): Patients assigned to the experimental group are included in an early occupational therapy intervention program.
  Interventions: Other: Early Occupational Therapy intervention
- Control group - Caregivers (No Intervention): Caregivers of patients who receive usual care and rehabilitation.
- OT intervention group - Caregivers (Experimental): Caregivers of the patients that are in the experimental group and are included in an early occupational therapy intervention program.
  Interventions: Other: Early Occupational Therapy intervention

INTERVENTIONS:
Other: Early Occupational Therapy intervention — four-week OT intervention program for patients who have suffered a stroke with the aim of improving the functional result and facilitating the return home by providing knowledge about specific care and neurorehabilitation.
  Arms: OT intervention group - Caregivers; OT intervention group - Patients

SUMMARY:
The general objective of this study is to determine if an early occupational therapy (OT) intervention together with the usual care at hospital discharge after suffering a stroke has a positive effect on the quality of life and functional independence of the patient, compared with the control group that will have the usual care and rehabilitation. We designed a four-week OT intervention program in patients who have suffered a stroke with the aim of improving the functional result and facilitating the return home by providing knowledge to the caregiver about specific care and neurorehabilitation.

DETAILED DESCRIPTION:
Background: Stroke is the leading cause of acquired disability in adults, being a cerebrovascular disease of great impact in health and social terms, due not only to its prevalence and incidence, but to the great repercussion in terms of dependence and its consequent impact on the life of the patient and family.

General and specific objectives: The general objective of this study is to determine if an early occupational therapy (OT) intervention together with the usual care at hospital discharge after suffering a stroke has a positive effect on the quality of life of the patient, compared with the control group that will have the usual care and rehabilitation. We designed a four-week OT intervention program with the support of the main caregiver in patients who have suffered a stroke with the aim of improving the functional result and facilitating the return home by providing knowledge about specific care and neurorehabilitation. Primary outcome: quality of life and functional independence. Secondary outcomes: improvement in sensory-motor skills, perceptual-cognitive skills, communication skills, levels of anxiety and depression of the patient, as well as caregivers' burden and coping strategies. The final results are evaluated three months after discharge.

Study Design: This is a prospective, randomized, controlled clinical trial. The sample size is made up of 60 patients who will be divided into two groups: the control group, with 30 users, and the experimental group, with another 30 users. The sample will be made up of patients who have suffered a stroke and have been discharged from the neurology service of a second-level hospital in West Malaga (Spain), being referred to the rehabilitation service by joint decision of the neurology and rehabilitation department. Patients assigned to the experimental group and their caregivers are included in an early occupational therapy intervention program and compared with a control group that receives usual care and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke with single or multiple vascular lesions that have occurred in the same time period, demonstrated by neuroimaging tests (CT or MRI).
* 18 years of age or older.
* Patient must live a maximum of 30 minutes away from the hospital center.
* Must present > 2 or <26 points on the National Institute of Health scale (NIHSS) and 30-100 points on the Barthel Index (BI) on the second day of the stroke (with BI 100, the patient can be included if the Montreal Cognitive Assessment is <26).
* Patient must present some motor deficit that makes it difficult to carry out his ADL.
* Inclusion in the study occurs prior to hospital discharge.

Exclusion Criteria:

* NIHSS> 26 and BI <30.
* Life expectancy <1 year.
* Previous stroke, dementia or other types of illnesses associated with dementia and other neurological, psychiatric or medical illnesses (for example, severe epilepsy, head trauma, schizophrenia, COPD, severe or unstable heart disease, sleep apnea) that could alter cognitive function.
* Moderate-severe aphasia.
* Does not understand Spanish or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PATRICIA GARCIA PEREZ, Principal Investigator — University of Malaga
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Perez P, Rodriguez-Martinez MC, Gallardo-Tur A, Blanco-Reina E, de la Cruz-Cosme C, Lara JP. Early Occupational Therapy Intervention post-stroke (EOTIPS): A randomized controlled trial. PLoS One. 2024 Aug 19;19(8):e0308800. doi: 10.1371/journal.pone.0308800. eCollection 2024. PMID 39159190

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of all the patients that were asked for enrollment, only 55 had a relative or friend as a caregiver and agreed to cooperate with the research.
Groups:
- Patients Control Group: Patients received usual care by ward and rehabilitation staff.
- Patients Experimental Group: EOTIPS Intervention.: Patients assigned to the experimental group are included in an early occupational therapy intervention program.
  Early Occupational Therapy intervention (EOTIPS): four-week OT intervention program with the support of the main caregiver in patients who have suffered a stroke with the aim of improving patient quality of life and facilitating the return home by providing knowledge to the caregiver about specific care and neurorehabilitation.
- Caregivers Control Group: Caregivers of patients who received usual care by ward and rehabilitation staff.
- Caregivers Experimental Group: Caregivers of patients assigned to the experimental group who are included in an early occupational therapy intervention program.
  Early Occupational Therapy intervention (EOTIPS): four-week OT intervention program with the support of the main caregiver in patients who have suffered a stroke with the aim of improving patient quality of life and facilitating the return home by providing knowledge to the caregiver about specific care and neurorehabilitation.
Period: Overall Study
Arm/Group | Patients Control Group | Patients Experimental Group: EOTIPS Intervention. | Caregivers Control Group | Caregivers Experimental Group
Started | 31 | 31 | 27 | 28
Completed | 30 | 30 | 27 | 28
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The sample size "n" was calculated to represent the total population of patients who suffer a stroke and are admitted to the Virgen de la Victoria University Hospital in Malaga, and who, after the neurological intervention, are left with sequelae susceptible to rehabilitation, but who do not acquire a place as inmates in the rehabilitation unit (a total of 800 stroke admissions to the Hospital are estimated per year).
Groups:
- Control Group - Patients: Usual care provided by hospital/community staff.
- EOTIPS (OT Intervention) - Patients: Patients and their caregivers assigned to the experimental group are included in an early occupational therapy intervention program.
  Early Occupational Therapy intervention: four-week OT intervention program with the support of the main caregiver in patients who have suffered a stroke with the aim of improving quality of life and facilitating the return home by providing knowledge to the caregiver about specific care and neurorehabilitation.
- Control Group - Caregivers: Caregivers of patients who received usual care by ward and rehabilitation staff.
- EOTIPS (OT Intervention) - Caregivers: Caregivers of patients assigned to the experimental group who are included in an early occupational therapy intervention program.
  Early Occupational Therapy intervention (EOTIPS): four-week OT intervention program with the support of the main caregiver in patients who have suffered a stroke with the aim of improving patient quality of life and facilitating the return home by providing knowledge to the caregiver about specific care and neurorehabilitation.
- Total: Total of all reporting groups
Arm/Group | Control Group - Patients | EOTIPS (OT Intervention) - Patients | Control Group - Caregivers | EOTIPS (OT Intervention) - Caregivers | Total
Number analyzed (Participants) | 31 | 31 | 27 | 28 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 24 | 23 | 81
  >=65 years | 15 | 13 | 3 | 5 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.6) | 68.5 (10.7) | 60 (22.3) | 61.2 (19.8) | 67.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 15 | 20 | 62
  Male | 16 | 19 | 12 | 8 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 25 | 25 | 23 | 101
  Not Hispanic or Latino | 3 | 6 | 2 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 31 | 31 | 27 | 28 | 117
Native language: spanish [Count of Participants; unit: Participants] | 29 | 29 | 26 | 26 | 110
Marital status [Count of Participants; unit: Participants] — Population: Caregivers were not assessed for this measure.
  Participants
    number analyzed (Participants) | 31 | 31 | 0 | 0 | 62
    Single | 2 | 3 |  |  | 5
    Divorced | 2 | 2 |  |  | 4
    Widowed | 6 | 6 |  |  | 12
    Married/living with partner | 21 | 20 |  |  | 41
Education [Count of Participants; unit: Participants] — Population: Caregivers were not assessed for this measure.
  Participants
    number analyzed (Participants) | 31 | 31 | 0 | 0 | 62
    No studies | 1 | 1 |  |  | 2
    Reads/writes | 8 | 12 |  |  | 20
    Primary school | 15 | 9 |  |  | 24
    High school | 5 | 3 |  |  | 8
    University | 2 | 6 |  |  | 8
Employment status [Count of Participants; unit: Participants] — Population: Caregivers were not assessed for this measure.
  Participants
    number analyzed (Participants) | 31 | 31 | 0 | 0 | 62
    Househusband/housewife | 1 | 4 |  |  | 5
    Unemployed | 2 | 1 |  |  | 3
    Retired | 20 | 18 |  |  | 38
    Temporary disability | 8 | 7 |  |  | 15
    Other activities | 0 | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Quality of Life
Description: Assessed with Stroke and aphasia quality of life scale-39 (SAQOL-39). Unit of measure will be the result of this assessment. Final score goes from 0 to 195 (higher score, better outcome).
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: Patients that enrolled EOTIPS program were assessed with SAQOL-39 in order to define wether their quality of life has improved, comparing to a control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group: Patients in control group received usual/standard care.
- OT Intervention.: Patients assigned to the experimental group are included in an early occupational therapy intervention program.
  Early Occupational Therapy intervention: four-week OT intervention program with the support of the main caregiver in patients who have suffered a stroke with the aim of improving the functional result and facilitating the return home by providing knowledge to the caregiver about specific care and neurorehabilitation.
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
score on a scale
  After intervention (3 months) | 3.41 (0.69) | 3.91 (0.70)
  Before intervention (baseline) | 2.51 (0.75) | 2.67 (0.72)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.029, ANOVA

2. Secondary Outcome: Patient's Sensory-motor Skills
Description: Assessed with Fugl Meyer Assessment (FMA). Unit of measure will be the result of this assessment. Total score is 0 to 126 (the higher score, the better upper limb sensory-motor skills).
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: All participants were assessed with Fugl-Meyer sensory motor assessment (FMA) in order to define wether EOTIPS program induced an improvement in the motor upper limb functions compared to the control group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
Score on a scale
  After intervention (3 months) | 111.10 (17.6) | 117 (12.6)
  Before intervention (baseline). | 99.80 (22.60) | 102.00 (18.90)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.148, ANOVA

3. Secondary Outcome: Patient Perceptual-cognitive Skills
Description: Assessed with Montreal Cognitive Assessment (MoCA). MoCA has been proposed as a screening tool that promises good sensitivity to deficits that result from stroke and vascular cognitive impairment. Unit of measure will be the result of this assessment.The final score goes from 0 to 30 (higher score, better outcome).
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: Cognitive impairment was assessed with Montreal Cognitive Assessment (MoCA) to define if cognition has improved in the EOTIPS group compared to the control group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
Score on a scale
  After intervention (3 months). | 20.1 (7.06) | 24.8 (6.58)
  Before intervention (baseline). | 16.6 (7.33) | 18.6 (7.16)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.012, ANOVA

4. Secondary Outcome: Patient Communication Skills
Description: Assessed with Communicative Activity Log (CAL). Scale that allows obtaining information on communication skills in activities of daily life referring to comprehensive and expressive aspects of language. Unit of measure will be the result of this assessment. Final score goes from 0 to 190 (higher score, better outcome).
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: Communication was assessed with Communicative Activity Log (CAL) to define if the communication skills were better in the EOTIPS group compared to the control group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
Score on a scale
  After intervention (3 months). | 116 (31.1) | 137 (24.2)
  Before intervention (baseline). | 109.00 (37.00) | 122.00 (27.30)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.078, ANOVA

5. Secondary Outcome: Depression of the Patient
Description: Assessed with Beck Depression Inventory (BDI-2). It is one of the most commonly used instruments to measure the severity of depression. Unit of measure will be the result of this assessment. Final score goes from 0 to 63 (lower score, better outcome).
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: Depression was assessed with Beck Depression Inventory (BDI-2) to define if the level of depression was lower in the EOTIPS group compared to the control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
score on a scale
  After intervention (3 months). | 15.3 (10.48) | 8.4 (8.88)
  Before intervention (baseline). | 13.60 (9.76) | 11.23 (9.11)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.011, ANOVA

6. Secondary Outcome: Patient Mobility
Description: Assessed with Time up and go (TUG). The TUG assesses basic mobility, timing the time required for a person to get up from a standardized chair, walk a distance of three meters, turn, return to the chair, and sit down again. Unit of measure will be the result of this assessment, which is the time in seconds. Shorter time means better performance.
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: Basic mobility was assessed with Timed Up and Go (TUG)) to define if it improved more in the EOTIPS group compared to the control group.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
seconds
  After intervention (3 months). | 12.4 (4.83) | 14.3 (12.8)
  Before intervention (baseline). | 28.40 (17.68) | 29.00 (12.90)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.797, ANOVA

7. Secondary Outcome: Patient Functional Balance
Description: Assessed with Berg Balance Scale (BBS) which evaluates assesses functional balance. Unit of measure will be the result of this assessment. Final score goes from 0 to 56 (higher score, better outcome).
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: Functional balance was assessed with Berg Balance Scale (BBS) to define if it improved more in the EOTIPS group compared to the control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
score on a scale
  After intervention (3 months). | 45.3 (11.7) | 47 (11.1)
  Before intervention (baseline). | 22.70 (17.90) | 27.60 (14.60)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.358, ANOVA

8. Secondary Outcome: Anxiety of the Patient
Description: Assessed with Hamilton anxiety scale. This scale assesses the severity of anxiety globally in patients who meet criteria for anxiety or depression. Unit of measure will be the result of this assessment. Final score goes from 0 to 56 (lower score, better outcome).
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: Anxiety of the patient was assessed with Hamilton anxiety scale to define if it improved more in the EOTIPS group compared to the control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
score on a scale
  After intervention (3 months). | 11.3 (9.4) | 5.5 (7.94)
  Before intervention (baseline). | 11.50 (10.88) | 8.47 (10.96)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.055, ANOVA

9. Secondary Outcome: Patient Functional Independence Assessed With Barthel Index
Description: The main unit of measure is the result of Barthel Index (from 0 to 100), 0 meaning disability and 100 meaning independence, therefore, higher score, better outcome. The main goal of this research is to assess independence of the patient and support needs in activities of daily living. The Barthel index measures the extent to which someone can function independently during basic activities of daily living.
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: The functional independence was assessed with Barthel Index to define if it improved more in the EOTIPS group compared to the control group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
score on a scale
  After intervention (3 months). | 85 (16.7) | 90 (14.9)
  Before intervention (baseline). | 52.5 (21) | 54.7 (20.5)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.496, ANOVA

10. Secondary Outcome: Patient Functional Independence Assessed With Stroke Impact Scale-16
Description: Unit of measure will be the result of this assessment. The score goes from 16 to 80, 80 meaning independence (higher score, better outcome). The usefulness of this scale is similar to that of the Barthel Index, although it is more sensitive than the latter to discriminate between patients with mild disabilities.
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: The functional independence was assessed with SIS-16 to define if it improved more in the EOTIPS group compared to the control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
score on a scale
  After intervention (3 months). | 61.9 (12.6) | 66.3 (10.7)
  Before intervention (baseline). | 36.60 (14.00) | 37.70 (11.00)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.241, ANOVA

11. Secondary Outcome: Patient Disability Assessed With Modified Rankin Scale (mRs)
Description: The mRS is used to describe disability in general. Unit of measure will be the result of this assessment. The score goes from 0 to 6, 0 meaning no symptoms and 6 meaning death (higher score, worse outcome).
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: The patient general disability was assessed with modified Rankin scale to define if it improved more in the EOTIPS group compared to the control group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group | OT Intervention.
Number analyzed (Participants) | 30 | 30
Score on a scale
  After intervention (3 months). | 2.5 (1.04) | 1.83 (1.05)
  Before intervention (baseline). | 3.60 (0.77) | 3.63 (0.80)
Statistical Analysis 1: Comparison: Control Group vs OT Intervention; Test type: Superiority; p = 0.004, ANOVA

12. Other Pre Specified Outcome: Caregiver Burden.
Description: Caregiver burden was evaluated with Caregiver Burden Scale (CBS). The Caregiver Burden Scale (CBS) is a 22-item scale that assesses the burden subjectively experienced by caregivers.The total score range is 0 to 88, where the higher the score, the more severe the burden: 0-21 no or mild burden, 21-40 mild to moderate burden, 41-60 moderate to severe burden, and ≥61 severe burden.
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: The caregivers that wanted to participate in the study were evaluated.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group - Caregivers | OT Intervention Group - Caregivers
Number analyzed (Participants) | 27 | 28
Score on a scale
  After intervention (3 months). | 3.91 (0.70) | 3.41 (0.69)
  Before intervention (baseline). | 12.8 (12.6) | 14.5 (6.91)
Statistical Analysis 1: Comparison: Control Group - Caregivers vs OT Intervention Group - Caregivers; Test type: Superiority; p = 0.019, ANOVA

13. Other Pre Specified Outcome: Caregivers Coping Strategies.
Description: The caregivers coping strategies were evaluated with the Coping Strategies Inventory (CSI), that was adapted to 40 items. The scale measures individual coping strategies that are broadly classified into two basic approaches to managing stressful situations: coping activities that involve the individual in the stressful situation (engagement strategies) and coping activities that disengage the individual (disengagement strategies). Total subscales score range are: disengagement strategies 0 to 60 and engagement strategies 0 to 60. The higher the score, the more strategies of that type they have.
Time Frame: Before intervention (baseline) and after intervention (3 months)
Population: The caregivers that were involved in the recovery of the patients were included in the study and evaluated.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group - Caregivers | OT Intervention Group - Caregivers
Number analyzed (Participants) | 27 | 28
Score on a scale
  Engagement strategies - BEFORE | 38.2 (12.6) | 42.5 (10.2)
  Disengagement strategies - BEFORE | 33.9 (6.8) | 36.4 (8.18)
  Engagement strategies - AFTER | 40.8 (13.6) | 49.0 (10.5)
  Disengagement strategies - AFTER | 37.4 (7.95) | 38.0 (7.6)
Statistical Analysis 1: Comparison: Control Group - Caregivers vs OT Intervention Group - Caregivers; ENGAGEMENT STRATEGIES; Test type: Superiority; p = 0.141, ANOVA
Statistical Analysis 2: Comparison: Control Group - Caregivers vs OT Intervention Group - Caregivers; DISENGAGEMENT STRATEGIES; Test type: Superiority; p = 0.496, ANOVA

ADVERSE EVENTS:
Time Frame: 18 months
Description: There were not adverse events reported.
Groups:
- Control Group - Patients: Participants that enroll control group received usual/standard care and rehabilitation.
- OT Intervention (EOTIPS) - Patients: Patients and their caregivers assigned to the experimental group are included in an early occupational therapy intervention program.
  Early Occupational Therapy intervention: four-week OT intervention program with the support of the main caregiver in patients who have suffered a stroke with the aim of improving the functional result and facilitating the return home by providing knowledge to the caregiver about specific care and neurorehabilitation.
- Control Group - Caregivers: Caregivers of the participants in the control group.
- OT Intervention (EOTIPS) - Caregivers: Caregivers of the participants in the experimental group.
Arm/Group | Control Group - Patients | OT Intervention (EOTIPS) - Patients | Control Group - Caregivers | OT Intervention (EOTIPS) - Caregivers
All-Cause Mortality (participants affected / at risk) | 1/31 | 1/31 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT04835363/Prot_SAP_000.pdf